CLINICAL TRIAL: NCT02161458
Title: Escitalopram Effects on CSF Amyloid Beta Total Concentrations
Brief Title: Escitalopram Effects on CSF Amyloid Beta
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01AG041502 (NIH)
Record Dates: First submitted 2014-06-05; First posted 2014-06-11 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Amyloid Beta Protein
Keywords: Escitalopram; Amyloid Beta; Cerebrospinal Fluid
MeSH Terms: conditions — Plaque, Amyloid | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Escitalopram 20mg for 2 weeks (Experimental): 30 cognitively normal adults aged 60-85 will receive escitalopram 20mg for 2 weeks (upward titration as: 10mg for 5 days, then 20mg for 9 days); and amyloid beta levels in the CSF will be measured at baseline (before drug administration) and after 2 weeks of study drug (active or placebo). Participants will taper off medication following the 2nd CSF measurement.
  Interventions: Drug: Escitalopram 20mg for 2 weeks
- Placebo (sugar pill) (Placebo Comparator): 30 cognitively normal adults aged 60-85 will receive placebo for 2 weeks (upward titration as: 10mg for 5 days, then 20mg for 9 days) or 8 weeks (upward titration as: 10mg for 5 days, then 20mg for 51 days); and amyloid beta levels in the CSF will be measured at baseline (before drug administration) and after 2 or 8 weeks of study drug (active or placebo). Participants will taper off medication following the 2nd CSF measurement.
  Interventions: Drug: Placebo
- Escitalopram 30mg for 8 weeks (Experimental): 30 cognitively normal adults aged 60-85 will receive escitalopram 30 mg for 8 weeks (upward titration as: 10mg for 5 days, then 20mg for 5 days; then 30 mg for 46 days); and amyloid beta levels in the CSF will be measured at baseline (before drug administration) and after 8 weeks of study drug (active or placebo). Participants will taper off medication following the 2nd CSF measurement.
  Interventions: Drug: Escitalopram 30mg for 8 weeks
- Escitalopram 20mg for 8 weeks (Experimental): 30 cognitively normal adults aged 60-85 will receive escitalopram 20mg for 8 weeks (upward titration as: 10mg for 5 days, then 20mg for 51 days); and amyloid beta levels in the CSF will be measured at baseline (before drug administration) and after 8 weeks of study drug (active or placebo). Participants will taper off medication following the 2nd CSF measurement.
  Interventions: Drug: Escitalopram 20mg for 8 weeks

INTERVENTIONS:
Drug: Escitalopram 20mg for 2 weeks — 30 cognitively normal adults aged 60-85 will receive escitalopram 20 mg for 2 weeks; amyloid beta levels in the CSF will be measured at baseline (before drug administration) and following the full study drug (i.e., active drug) administration.
  Arms: Escitalopram 20mg for 2 weeks
Drug: Escitalopram 20mg for 8 weeks — 30 cognitively normal adults aged 60-85 will receive escitalopram 20 mg for 8 weeks; amyloid beta levels in the CSF will be measured at baseline (before drug administration) and following the full study drug (i.e., active drug) administration.
  Arms: Escitalopram 20mg for 8 weeks
Drug: Escitalopram 30mg for 8 weeks — 30 cognitively normal adults aged 60-85 will receive escitalopram 30 mg for 8 weeks; amyloid beta levels in the CSF will be measured at baseline (before drug administration) and following the full study drug (i.e., active drug) administration.
  Arms: Escitalopram 30mg for 8 weeks
Drug: Placebo — Additionally, 30 cognitively normal adults aged 60-85 will receive a placebo; amyloid beta levels in the CSF will be measured at baseline (before drug administration) and following the full study drug (i.e., placebo) administration.
  Arms: Placebo (sugar pill)

SUMMARY:
Alzheimers disease (AD) is a devastating illness, estimated to affect 5 million patients in the United States alone and projected to increase dramatically over the next decades as the population ages unless preventive measures can be developed. The investigators have preliminary evidence that selective serotonin reuptake inhibitor (SSRI) antidepressants lower the amount of amyloid plaques in the human brain. The interventions now propose to study the effects of an SSRI (escitalopram) on levels of amyloid beta peptide (the major constituent of the plaques) in the cerebrospinal fluid (CSF) of cognitively normal older adults.

DETAILED DESCRIPTION:
The investigators will measure CSF Amyloid Beta levels before and after two weeks or eight weeks of treatment with escitalopram using a double blind placebo-controlled study design with approximately 30 cognitively normal participants, age 60-85, with a MOCA of 23 or higher. They will be recruited from the community. Participants will be randomized (approximately 30 per group).

Participants in the 2 week arm will have 3 study visits:

1. Screening Visit: Consent and screening procedures will be complete. Participants will be randomized 1:1 to receive escitalopram or placebo.
2. Study Visit 1: This visit will take approximately 45 minutes - 1 hour; participants will have a lumbar puncture (LP) in order to obtain cerebrospinal fluid (CSF), a blood draw, and will receive study medication.
3. Study Visit 2: This visit will take approximately 45 minutes - 1 hour; participants will have a lumbar puncture (LP) in order to obtain cerebrospinal fluid (CSF), a blood draw, will receive taper-down study medication, and will complete an end-of-study questionnaire.

Participants in the 8-week arm(s) will have 4 study visits:

1. Screening Visit: Consent and screening procedures will be complete. Participants will be randomized 1:1 to receive escitalopram or placebo.
2. Study Visit 1: This visit will take approximately 45 minutes - 1 hour; participants will have a lumbar puncture (LP) in order to obtain cerebrospinal fluid (CSF), a blood draw, and will receive 4 weeks of study medication.
3. Study Visit 2: Researchers will check in with participants and participants will receive another 4 weeks of study medication.
4. Study Visit 3:This visit will take approximately 45 minutes - 1 hour; participants will have a lumbar puncture (LP) in order to obtain cerebrospinal fluid (CSF), a blood draw, will receive taper-down study medication, and will complete an end-of-study questionnaire.

The current proposal will test whether clinically relevant doses of an SSRI reduce CSF levels of Amyloid Beta in healthy older human participants. The investigators hypothesize that compared to placebo, participants receiving escitalopram will show significantly lower Amyloid Beta levels in the second CSF sample.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 60-85 (inclusive), male and female, any race.
* 2) Capacity to give informed consent and follow study procedures.
* 3) English speaking.
* 4) MOCA = 23 or greater

Exclusion Criteria:

* 1) Known history of relevant severe drug allergy or hypersensitivity (e.g. to Citalopram or Escitalopram)
* 2) Does not speak English
* 3) Cannot give informed consent
* 4) Diagnosis of Major Depression
* 5) Previous history of neurological disorders, such as Parkinson's disease, Alzheimer's disease or traumatic brain injury, cognitive impairment or dementia.
* 6) Diagnosis of a chronic psychiatric illness
* 7) Significant hearing or visual impairment
* 8) Bleeding diathesis
* 9) Clinically significant hepatic, renal, pulmonary, metabolic or endocrine disturbances as indicated by history, which in the opinion of the investigator might pose a potential safety risk to the subject.
* 10) Current clinically significant cardiovascular disease. Clinically significant cardiovascular disease usually includes one or more of the following: cardiac surgery or myocardial infarction within the last 4 weeks; unstable angina; acute decompensated congestive heart failure or class IV heart failure; current significant cardiac arrhythmia or conduction disturbance, particularly those resulting in ventricular fibrillation, or causing syncope or near syncope; uncontrolled high blood pressure; QTc greater than 450msec (by history for subjects with cardiac disease); documented prior stroke.
* 11) Clinically significant abnormalities on EKG. Primary AV block or Right bundle branch block are not necessarily exclusionary.
* 12) History of drug or alcohol abuse within the last year or prior prolonged history of abuse
* 13) Use of an Investigational medicine within the past 30 days 14) Use of Coumadin, Warfarin or other blood thinners within the past 6 months
* 15) Use of antipsychotic medication or antidepressant medication (e.g. MAOIs, SSRIs, SNRIs).
* 16) Use of the following drug/drug classes: Pimozide, Triptans, Tricyclics, Lithium, Tramadol
* 17) Use of over-the-counter supplements such as tryptophan or St. Johns Wort 18) Any other factor that in the investigator's judgment may affect patient safety or compliance (e.g. distance greater than 100 miles from the research institution)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-06; Primary Completion 2017-08 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Sheline, M.D., Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Washington University, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheline YI, Snider BJ, Beer JC, Seok D, Fagan AM, Suckow RF, Lee JM, Waligorska T, Korecka M, Aselcioglu I, Morris JC, Shaw LM, Cirrito JR. Effect of escitalopram dose and treatment duration on CSF Abeta levels in healthy older adults: A controlled clinical trial. Neurology. 2020 Nov 10;95(19):e2658-e2665. doi: 10.1212/WNL.0000000000010725. Epub 2020 Sep 10. PMID 32913021

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Escitalopram 20mg for 2 Weeks | Placebo (Sugar Pill) | Escitalopram 30mg for 8 Weeks | Escitalopram 20mg for 8 Weeks
Started | 22 | 35 | 33 | 8
Completed | 22 | 29 | 28 | 8
Not Completed | 0 | 6 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 4 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram 20mg for 2 Weeks | Placebo (Sugar Pill) | Escitalopram 30mg for 8 Weeks | Escitalopram 20mg for 8 Weeks | Total
Number analyzed (Participants) | 22 | 29 | 28 | 8 | 87
Age, Continuous [Mean (Full Range); unit: years] | 71 [60 to 79] | 70 [59 to 83] | 67 [60 to 78] | 65 [60 to 70] | 69 [59 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 14 | 5 | 36
  Male | 14 | 20 | 14 | 3 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 4 | 1 | 13
  White | 17 | 24 | 24 | 7 | 72
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 29 | 28 | 8 | 87

OUTCOME MEASURES:

1. Primary Outcome: Amyloid Beta Levels in CSF
Description: Change in the level of Amyloid Beta peptides (Amyloid Beta 42 and Amyloid Beta 40) in the CSF between the measurement at baseline and the measurement after exposure with escitalopram.
Time Frame: 2 - 8 Weeks (we used week 8 minus baseline and week 2 minus baseline)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Escitalopram 20mg for 2 Weeks | Placebo (Sugar Pill) | Escitalopram 30mg for 8 Weeks | Escitalopram 20mg for 8 Weeks
Number analyzed (Participants) | 22 | 29 | 28 | 8
pg/mL
  Ab 42 in CSF | -12.7 (24.43) | 6.74 (45.16) | -22.73 (43.80) | -25.63 (23.29)
  Ab 40 in CSF | 46.27 (539.29) | 197.36 (540.82) | -152.64 (572.90) | -41.82 (1039.83)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for up to 2 weeks after participants were active in the study, from the time of consent to the participant's last study visit.
Arm/Group | Escitalopram 20mg for 2 Weeks | Placebo (Sugar Pill) | Escitalopram 30mg for 8 Weeks | Escitalopram 20mg for 8 Weeks
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/29 | 0/28 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/29 | 0/28 | 0/8
Other Adverse Events (participants affected / at risk) | 0/22 | 0/29 | 0/28 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT02161458/Prot_SAP_001.pdf